CLINICAL TRIAL: NCT00281554
Title: A Phase 3, Multi-Center, Open Label, Safety Study of RSD1235 in Subjects With Atrial Fibrillation
Brief Title: Study of RSD1235 to Evaluate Safety in Patients With Atrial Fibrillation
Acronym: ACT 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Advanz Pharma (Industry)
Responsible Party: Sr Manager Clinical Trial Registry, Astellas Pharma US, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-7-012
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Atrial Fibrillation
Keywords: Investigational Therapies; Atrial Fibrillation; Treatment Efficacy; Treatment Effectiveness; Safety; RSD1235
MeSH Terms: conditions — Atrial Fibrillation | interventions — vernakalant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RSD1235

INTERVENTIONS:
Drug: RSD1235 — IV
  Other Names: vernakalant; Kynapid

SUMMARY:
This study is designed to determine the safety of RSD1235 in patients with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have symptomatic AF
* Subject must have adequate anticoagulant therapy

Exclusion Criteria:

* Subject may not have Class IV congestive heart failure.
* Subject may not have uncorrected electrolyte imbalance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2005-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Rate of conversion of atrial fibrillation to sinus rhythm for a minimum of 1 minute | Infusion plus 1.5 hours

SECONDARY OUTCOMES:
Evaluate safety | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (35):
- United States (10):
  - Huntsville, Alabama
  - Atlanta, Georgia
  - Chicago, Illinois
  - Oak Lawn, Illinois
  - Boston, Massachusetts
  - Lansing, Michigan
  - Austin, Texas
  - San Antonio, Texas
  - Richmond, Virginia
  - Marshfield, Wisconsin
- Argentina (5):
  - Buenos Aires
  - Corrientes
  - De Buenos Aires
  - Rosario
  - Tulunaw
- Canada (4):
  - Calgary, Alberta
  - Ottawa, Ontario
  - Montreal, Quebec
  - Terrebonne, Quebec
- Denmark (6):
  - Aalborg
  - Esbjerg
  - Hjørring
  - Hvidovre
  - København NV
  - Køge
- South Africa (6):
  - Berea Durban
  - Bloemfontein
  - Centurion
  - Parow
  - Somerset West
  - Westdene Bloemfontein
- Sweden (4):
  - Malmo
  - Mölndal
  - Örebro
  - Stockholm

REFERENCES:
- [Derived] Stiell IG, Dickinson G, Butterfield NN, Clement CM, Perry JJ, Vaillancourt C, Calder LA. Vernakalant hydrochloride: A novel atrial-selective agent for the cardioversion of recent-onset atrial fibrillation in the emergency department. Acad Emerg Med. 2010 Nov;17(11):1175-82. doi: 10.1111/j.1553-2712.2010.00915.x. PMID 21175515
- [Derived] Stiell IG, Roos JS, Kavanagh KM, Dickinson G. A multicenter, open-label study of vernakalant for the conversion of atrial fibrillation to sinus rhythm. Am Heart J. 2010 Jun;159(6):1095-101. doi: 10.1016/j.ahj.2010.02.035. PMID 20569725